CLINICAL TRIAL: NCT04769362
Title: Discontinuation of β-blocker Therapy in Stabilized Patients After Acute Myocardial Infarction: A Multicenter Randomized Noninferiority Trial
Brief Title: Long-term Beta-blocker Therapy After Acute Myocardial Infarction
Acronym: SMART-DECISION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Gyeongsang National University Hospital (Other); Kyung Hee University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Sejong General Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Changwon Hospital (Other); Saint Vincent's Hospital, Korea (Other); Presbyterian medical center (Unknown); Wonkwang University Hospital (Other); Wonju Severance Christian Hospital (Other); Ewha Womans University Seoul Hospital (Other); Inje University Ilsan Paik Hospital (Other); Chonbuk National University Hospital (Other); Chonnam National University Hospital (Other); Jeju National University Hospital (Other); Chosun University Hospital (Other); Chungbuk National University Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, MD, PhD, Division of Cardiology, Department of Medicine, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC202010176
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-blocker discontinuation arm (Experimental): Discontinuation of β-blocker therapy after at least 1 year of β-blocker therapy after acute myocardial infarction
  Interventions: Drug: Discontinuation of β-blocker
- β-blocker maintenance arm (No Intervention): Continuation of β-blocker therapy after acute myocardial infarction

INTERVENTIONS:
Drug: Discontinuation of β-blocker — Discontinuation of β-blocker after at least 1 year of β-blocker therapy after acute myocardial infarction
  Arms: β-blocker discontinuation arm

SUMMARY:
The aim of the study is to determine whether discontinuation of β-blocker after at least 1 year of β-blocker therapy is noninferior to continuation of β-blocker in patients without heart failure (HF) or left ventricular systolic dysfunction after acute myocardial infarction (AMI).

Prospective, open-label, randomized, multicenter, noninferiority trial to determine whether discontinuation of β-blocker after at least 1 year of β-blocker therapy is noninferior to continuation of β-blocker in patients without HF or left ventricular systolic dysfunction after AMI.

DETAILED DESCRIPTION:
β-blockers have anti-ischemic, anti-arrhythmic, and anti-adrenergic properties. In order to reduce cardiovascular mortality and morbidity, current major guidelines recommend that oral treatment of β-blockers should be continued during and after hospitalization in patients with acute myocardial infarction (AMI) and without contraindications to β-blocker use.

A clinically important but difficult decision on β-blocker therapy after AMI is to determine the duration of β-blocker therapy after discharge in patients without heart failure (HF) or left ventricular systolic dysfunction. Previous studies for long-term β-blocker therapy after AMI were inadequate to derive definite conclusion because of small sample size and potential selection bias.

Therefore, the SMART-DECISION trial will investigate whether discontinuation of β-blocker after at least 1 year of β-blocker therapy is noninferior to continuation of β-blocker in patients without HF or left ventricular systolic dysfunction after AMI.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age.
* Subject who have been continuing β-blocker therapy for at least 1 year after acute myocardial infarction regardless of the time of diagnosis
* Subject is able to verbally confirm understandings of risks and benefits of this trial, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Subject whose left ventricle ejection fraction was less than 40% from echocardiography performed after acute myocardial infarction or who have never received echocardiography.
* Treatment history of heart failure
* Contraindication to β-blocker therapy (history of symptomatic bronchial asthma or chronic obstructive pulmonary disease, 2nd or 3rd degree AV block, cardiac pacemaker implantation, or other cases where β-blocker cannot be used under the judgment of the clinician)
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* History of atrial fibrillation
* Pregnancy or breast feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2540 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 2.5 years after last patient enrollment
  a composite of all-cause death, myocardial infarction, hospitalization for heart failure

SECONDARY OUTCOMES:
All-cause death | 2.5 years after last patient enrollment
Cardiovascular death | 2.5 years after last patient enrollment
Myocardial infarction | 2.5 years after last patient enrollment
Any hospitalization | 2.5 years after last patient enrollment
Hospitalization for heart failure | 2.5 years after last patient enrollment
Hospitalization for acute coronary syndrome | 2.5 years after last patient enrollment
All-cause death or myocardial infarction | 2.5 years after last patient enrollment
Cardiovascular death or myocardial infarction | 2.5 years after last patient enrollment
Myocardial infarction or hospitalization for heart failure | 2.5 years after last patient enrollment
Any revascularization | 2.5 years after last patient enrollment
Myocardial infarction or any revascularization | 2.5 years after last patient enrollment
Cardiovascular death, myocardial infarction, or hospitalization for heart failure | 2.5 years after last patient enrollment
Cardiovascular death, myocardial infarction, or any revascularization | 2.5 years after last patient enrollment
left ventricle ejection fraction | at 2 years
  changes in left ventricle ejection fraction
N-terminal pro-brain natriuretic peptide (NT-proBNP) | 2.5 years after last patient enrollment
  changes in NT-proBNP
Atrial fibrillation occurrence | 2.5 years after last patient enrollment
Medical cost | at 2 years
  The medical expenses related to heart problems during the follow-up
PROMIS 29 | 2.5 years after last patient enrollment
  PROMIS 29 is composed of a total of 29 questions, and questions are composed of domains for physical function, anxiety, depression, sleep, social function, participation availability, and pain.
Adverse effects related with β-blocker | 2.5 years after last patient enrollment
Rate of Hospitalization for cardiovascular causes | 2.5 years after last patient enrollment
  Rate of Hospitalization for cardiovascular causes
Rate of Stroke | 2.5 years after last patient enrollment
  Rate of ischemic or hemorrhagic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD,PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.

REFERENCES:
- [Derived] Choi KH, Kim J, Kang D, Doh JH, Kim J, Park YH, Ahn SG, Kim W, Park JP, Kim SM, Cho BR, Nam CW, Cho JH, Joo SJ, Suh J, Jeong JO, Jang W, Yoon CH, Hwang JY, Lim SH, Lee SR, Shin ES, Kim BJ, Yu CW, Her SH, Kim HK, Park KT, Kim J, Park TK, Lee JM, Cho J, Yang JH, Song YB, Choi SH, Gwon HC, Guallar E, Hahn JY; SMART-DECISION investigators. Discontinuation of beta-blocker therapy in stabilised patients after acute myocardial infarction (SMART-DECISION): rationale and design of the randomised controlled trial. BMJ Open. 2024 Aug 31;14(8):e086971. doi: 10.1136/bmjopen-2024-086971. PMID 39645270